CLINICAL TRIAL: NCT02838082
Title: Optimized Sleep After Brain Injury: A Pilot Study
Brief Title: Optimized Sleep After Brain Injury: Sleep Hygiene Intervention After Traumatic Brain Injury
Acronym: OSABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: Colorado Traumatic Brain Injury Trust Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 839979IRB
Record Dates: First submitted 2016-06-24; First posted 2016-07-20 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; sleep-wake cycle disturbance; circadian disruption
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

ARMS (2):
- Sleep Hygiene Protocol (Experimental): Participants in this arm will undergo a 4 week sleep hygiene protocol
  Interventions: Behavioral: Sleep Hygiene Protocol
- Standard of Care Protocol (Active Comparator): Participants will undergo 4 weeks of current inpatient standard of care procedures in a rehabilitation facility
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Sleep Hygiene Protocol — Sleep Hygiene Protocol involving 1) Improved sleep environment 2) Enhanced Circadian Stimuli 3) Increased Daytime Activation (blue light therapy, daytime light exposure and daytime sleep restriction) 4) Adjusted morning ADL routines and 5) Restricted Caffeine intake
  Arms: Sleep Hygiene Protocol
Behavioral: Standard of Care — All standard of care procedures in a specialized traumatic brain injury inpatient rehabilitation unit
  Arms: Standard of Care Protocol

SUMMARY:
OSABI is a pilot study of a sleep hygiene protocol for sleep disruptions associated with TBI during inpatient rehabilitation. Twenty participants will be allocated (by minimization) either into a standard of care protocol or a sleep hygiene protocol for 4 weeks. Sleep efficiency (via actigraphy), post traumatic amnesia (OLOG), agitation (Agitated Behavior Scale) and cognitive function (Confusion Assessment Protocol) will be monitored during the trial period to examine relationships among them.

DETAILED DESCRIPTION:
Estimates of sleep disruption after traumatic brain injury (TBI) reach 81%, but the incidence nature, course and effect on recovery from TBI are not well understood because most TBI sleep studies included mixed TBI severity samples at varied times post injury. In the early rehabilitation phase of recovery from moderate-to-severe TBI, sleep disturbance has been estimated at 78% and has been associated with the presence of post-traumatic amnesia (PTA); a transient period of disorientation, confusion and inability to store memories that occurs after TBI. Individuals with TBI who are in PTA not only have severe memory dysfunction that significantly impairs their ability to benefit from verbal instruction, but are often in a confusional state with agitated behavior. They require a 24-hour, highly structured environment for safety until their PTA resolves. PTA can last from days to weeks, during which time the individual and his/her family are significantly distressed. Its duration also has practical implications in terms of resources, length of hospitalization and cost.

There appears to be a relationship between sleep disturbance and PTA during early recovery from TBI, but the nature of the relationship is not fully understood. Sleep disturbance has been associated with delirium in non-TBI medical patients, and sleep deprivation has been associated with significant negative effects on attention, reaction time, visual-motor performance, language functions, memory processes, and executive functions in normal populations. Sleep disturbance appears to negatively affect cognitive functioning in both medical and normal samples. In the TBI population, sleep disruption could further exacerbate the already compromised cognitive functions and prolong PTA. The relationship between sleep disruption and PTA presents a potentially significant therapeutic opportunity because PTA is largely considered to be fixed and immutable with no therapeutic options. Therapeutic efforts to improve sleep may reduce the length of PTA.

The proposed study will begin to address the gap in knowledge about the nature, incidence and effect of sleep disturbances on recovery from moderate-to-severe TBI during the early rehabilitation period. It will also pilot a sleep hygiene protocol to improve sleep for individuals in the early rehabilitation phase after TBI. It will employ 24-hour per day sleep observations and actigraphy to characterize the incidence and type of sleep disturbances in the early rehabilitation phase of TBI. In addition, the study will serially test participants multiple times a week with the Orientation Log (OLOG) and the Confusion Assessment Protocol (CAP) to closely monitor changes in alertness, orientation, attention, memory functions and behavior as they emerge from PTA. The sleep observations and actigraph information can then be compared to the cognitive measures of PTA to examine the relationship of sleep quantity and quality on cognitive functions during recovery from PTA.

The randomized controlled trial with minimization allocation (RCT) pilot component of the study will be the first therapeutic attempt that we are aware of; to normalize sleep cycles and sleep quality in individuals with TBI who have sleep disruptions during early rehabilitation. Twenty individuals with TBI who have low sleep efficiency on actigraphy during the initial night time screening will be randomized into a comprehensive sleep hygiene protocol (SHP = 10) or a standard of care (SOC = 10) protocol for three weeks. Both groups will have access to all rehabilitation facilities, therapies, services and programs. The difference between the groups is the systematic attempt to improve sleep in the SHP by five principle components: 1) improved night sleep environment, 2) increased daytime activation, 3) enhanced circadian stimuli, 4) morning ADL routines individually adjusted to pre-injury biological sleep patterns and 5) no caffeine intake. In the SOC group, there will be no systematic efforts to influence circadian rhythms, daytime activation or nighttime sleep environment. Participant's sleep in both groups will be monitored with 24-hour actigraphy and staff ratings of sleep-awake periods throughout the 24 hour period on the Makley Sleep Scale (MSS) for four weeks. Additionally, nursing staff will rate agitation on the Agitated Behavior Scale and therapy staff will monitor cognitive functioning with the Orientation Log (OLOG) and Confusion Assessment Protocol (CAP) until after emergence from PTA. The sleep data, cognitive testing and behavioral information for both groups will enable examination of the relationship of sleep to PTA and the potential benefit of the SHP on normalizing sleep and enhancing cognitive recovery, including resolution of PTA.

ELIGIBILITY:
Inclusion Criteria:

* All male inpatient admissions to Craig Hospital with the primary diagnosis of TBI
* Rancho Level of Cognitive Functioning Scale >= III
* Ages >= 18 and < =55
* Fluent in the English language
* Available upper extremity for actigraph placement
* Average sleep efficiency= < 75 for three consecutive nights as measured by clinical actigraphy
* Physician judgment that the individual is in post-traumatic amnesia

Exclusion Criteria:

* Medical conditions that require intensive nursing care during the night time sleep period as determined by physician, e.g. tracheostomy
* Hydrocephalus with V-P shunt
* Penetrating Head Injury
* Anoxia associated with TBI
* Stroke associated with TBI
* Spinal cord injury associated with TBI
* Halo Fixation for cervical spine fracture
* Greater than 90 days post injury on admission to Craig Hospital
* Out of Post Traumatic Amnesia on screening
* Severe agitation that would make participation in the study unsafe as determined by the attending physician
* Unable to complete verbal assessments
* History of previous TBI requiring hospitalization
* History of neurodegenerative disease or dementing illness
* History of pre-existing diabetes, pre-disposing factors for diabetes
* History of retinal disease
* History of pre-existing diagnosis of Schizophrenia or Bi-Polar Disorder
* History of Active Major Depressive Illness prior to injury
* History of a diagnosed sleep disorder per family report or medical history
* History of Sleep Disordered Breathing such as sleep apnea as determined by history obtained from significant other/family member or medical history
* History of night shift work or of not being in a consistently standard sleep wake schedule during three months prior to TBI as determined by history obtained from significant other/family member or medical history.
* History of untreated/uncontrolled thyroid disease
* Individuals with epilepsy
* Individuals with central or peripheral blindness
* Body mass index greater than 30.
* Enrollment in a concurrent interventional clinical trial
* Estimated length of stay < 4 weeks
* Medical Proxy unavailable to consent

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Actiwatch Sleep Efficiency | 4 weeks
  Sleep efficiency via actigraphy is recorded nightly for 4 weeks

SECONDARY OUTCOMES:
Agitated Behavior Scale | 4 weeks
  Nursing staff ratings on the Agitated Behavior Scale each shift
Makley Sleep Scale | 4 weeks
  Staff observations/ratings of sleep every two hours
Orientation Log (O-Log) | 4 weeks
  Speech Pathology assessment of post traumatic amnesia with the O-Log 5 days per week
Confusion Assessment Protocol (CAP) | 4 weeks
  Neuropsychology Assessment of cognitive status with the CAP three days per week

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

REFERENCES:
- [Derived] Makley MJ, Gerber D, Newman JK, Philippus A, Monden KR, Biggs J, Spier E, Tarwater P, Weintraub A. Optimized Sleep After Brain Injury (OSABI): A Pilot Study of a Sleep Hygiene Intervention for Individuals With Moderate to Severe Traumatic Brain Injury. Neurorehabil Neural Repair. 2020 Feb;34(2):111-121. doi: 10.1177/1545968319895478. Epub 2019 Dec 30. PMID 31884895
- [Derived] Draganich C, Gerber D, Monden KR, Newman J, Weintraub A, Biggs J, Philippus A, Makley M. Disrupted sleep predicts next day agitation following moderate to severe brain injury. Brain Inj. 2019;33(9):1194-1199. doi: 10.1080/02699052.2019.1631484. Epub 2019 Jun 19. PMID 31215813